CLINICAL TRIAL: NCT02732613
Title: Selection of Laryngeal Mask Airway When Actual Body Weight Much Less Than Ideal Body Weight in Adult Patients
Brief Title: Selection of Laryngeal Mask Airway in Patients With Slender Somatotype
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: XiQiang Huang (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor-Investigator, XiQiang Huang, Attending doctor, Department of anesthesiology, Principal Investigator, Zhongshan People's Hospital, Guangdong, China
Organization: Zhongshan People's Hospital, Guangdong, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: ZSPH20160303
Record Dates: First submitted 2016-03-28; First posted 2016-04-08 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Size of Laryngeal Mask Airway; Body Weight; Success Rate of First Attempt; Complication
Keywords: Laryngeal Mask Airway; Body weight; Complication
MeSH Terms: conditions — Body Weight | interventions — Laryngeal Masks

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Actual weight Group (Experimental): Patients in Actual weight Group: The selection of Laryngeal Mask Airway classic will be based on actual body weight, followed the recommendations of manufacturer (size 3 for weight < 50 kg, size 4 for weight 50-70 kg, and size 5 for weight > 70 kg ).
  Interventions: Device: Laryngeal Mask Airway
- Ideal weight Group (Experimental): Patients in Ideal weight Group: The selection of Laryngeal Mask Airway classic will be based on ideal body weight, followed the recommendations of manufacturer ( size 3 for weight < 50 kg, size 4 for weight 50-70 kg, and size 5 for weight > 70 kg ).
  Interventions: Device: Laryngeal Mask Airway

INTERVENTIONS:
Device: Laryngeal Mask Airway — If there were any conflicts of the Laryngeal Mask Airway classic size selection in slim patients by the actual or ideal body weight, size selection will based on actual body weight in Actual weight Group while ideal body weight in Ideal weight Group.

SUMMARY:
The size selection of Laryngeal Mask Airway classic is usually followed the manufacturer's recommendation based on the patient's ideal weight. But sometimes the patient is tall and slim, the actual weight is much less than the ideal weight. This phenomenon might affect the success rate of insertion. Previous studies had demonstrated that the selection of Laryngeal Mask Airway size based on ideal weight could improve the success rate of insertion; therefore, this study was designed to prove whether this conclusion also applies to the tall and thin patients.

DETAILED DESCRIPTION:
One hundred and eighteen patients adult patients，actual body weight much less than ideal body weight will be assigned randomly to two groups (Actual weight Group or Ideal weight Group). Size selection was guided by the recommendations of manufacturer, patients will be based on the actual body weight in Actual weight Group while ideal body weight in Ideal weight Group.

The success rate of first attempt，number of adjustments, insertion time, ease of insertion, overall success rate, oropharyngeal leak pressure and fiberoptic view will be recorded and compared. The occurrences of respiratory complications such as sore throat, hoarseness, and dysphonia will be observed and recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Patients undergo elective surgery of American Society of Anesthesiologists (ASA) physical status 1-2, aged from 18 to 60;
2. Patients' actual weight much less than ideal weight.

Exclusion Criteria:

1. Patients with gastroesophageal reflux disease;
2. Patients with predicted difficult airway;
3. Patients with preexisting airway diseases or significant upper airway infection.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 118 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-09 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
The success rate of Laryngeal Mask Airway first insertion | Six months

IPD SHARING:
Plan to Share IPD: Undecided